CLINICAL TRIAL: NCT07355660
Title: The Effect of a Web-Based Education Program on Eating Habits, Metabolic Control, and Self-Management in Adolescents With Type 1 Diabetes Mellitus and Their Mothers With Irregular Eating Behavior
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Scientific and Technological Research Council of Turkey (Unknown)
Responsible Party: Principal Investigator, Gökhan GÖNÜL, Lecturer, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ERU-SBF-GG-01
Record Dates: First submitted 2026-01-06; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: In the first phase of the study, adolescents with disordered eating behaviors will be identified by administering the Descriptive Characteristics and Disordered Eating Behavior Scale (DESPR) to adolescents and their mothers. The sample for this phase was determined to be 272 adolescents using the G Power program with a d=0.2, a 0.05 margin of error, and a 95% confidence interval. For the second phase, adolescents with a DESPR score of 20 or higher will be divided into three groups: Intervention I (Adolescents Only), Intervention II (Adolescents and Their Mothers), and the Control Group (Clinical Practice Routine). The G Power program calculated that 24 individuals would be included in each group. This study will employ a block-randomized pretest-posttest design. The experimental group will receive a web-based education program, while the control group will receive only standard education and routine care.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group I (Adolescents) (Active Comparator)
  Interventions: Behavioral: Eating habits, Diabetes self-management, Metabolic control
- Intervention Group II (Adolescents and Their Mothers) (Active Comparator)
  Interventions: Behavioral: Eating habits, Diabetes self-management, Metabolic control
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Eating habits, Diabetes self-management, Metabolic control — This study addresses these gaps and offers a unique approach. Initially, unlike existing studies, the goal is to develop a holistic educational model encompassing both adolescents and their mothers. Furthermore, the program will be structured with content specific to disordered eating behaviors, which frequently coexist with Type 1 diabetes. In this respect, the project is one of the few initiatives that address the relationship between eating disorders and metabolic control in a holistic manner. Furthermore, the study is not limited to knowledge or self-management, but conducts a multidimensional analysis by jointly evaluating eating habits, metabolic parameters, and psychosocial indicators. The web-based content will be designed to suit the Turkish cultural context and will also allow for the assessment of the impact of variables such as digital inequality and parental support.
  Arms: Intervention Group I (Adolescents); Intervention Group II (Adolescents and Their Mothers)

SUMMARY:
The study was planned as a randomized controlled experimental study to investigate the effects of a web-based educational program given to adolescents with diabetes mellitus and their mothers on eating habits, metabolic control, and self-management.

The prevalence of Type 1 diabetes is increasing worldwide and is reported to be the third most common chronic disease in childhood (Lowes et al., 2015). It is generally accepted that effective management of diabetes requires education for both the patient and the family regarding management components such as blood glucose monitoring, insulin replacement, diet, exercise, and problem-solving strategies (Couch et al., 2008). Since diabetes management requires lifestyle changes, many health professionals recommend providing education to the whole family (Shiel et al., 2023).

Adolescence is a period of developing autonomy and often means reduced parental involvement; however, an adolescent with Type 1 diabetes is also coping with a serious, life-threatening disease (Polfuss et al., 2015). Increased self-care responsibilities during adolescence create additional complex challenges for the management and treatment of diabetes. Websites providing information about diabetes to adolescents offer problem-solving opportunities and an interactive environment for sharing experiences.

The study population will consist of adolescents and their mothers followed at the Pediatric Endocrinology Outpatient Clinic of Erciyes University Mustafa Eraslan and Fevzi Mercan Children's Hospital. In the first phase of the study, the Descriptive Characteristics and Eating Disorder Behavior Scale (DESPR) will be administered to adolescents and their mothers to identify adolescents with eating disorder behaviors. The sample was determined as 272 adolescents using the G Power program with a margin of error of d=0.2, a margin of error of 0.05, and a 95% confidence interval. For the second phase of the study, adolescents with a DESPR score of 20 or higher will be divided into three groups: Intervention I (Adolescents Only), Intervention II (Adolescents and Mothers), and Control Group (Clinical Practice Routine). The sample size was calculated using the G Power program with a margin of error of d=0.4, a margin of error of 0.05, and an 85% confidence interval, resulting in a total of 72 individuals, with 24 individuals in each group. The groups into which individuals will be placed will be determined using the block randomization method applied on the www.randomizer.org website.

Training Implementation:

Training will be given to two groups: Web-Based Intervention Group I (Adolescents) and Intervention Group II (Adolescents and Mothers). An initial introductory meeting will be held, and training on how to use the web program will be given in a single 40-minute session. Website Preparation: The website will be structured using WordPress, a web-based software development tool that supports most web browsers. Website content will be evaluated using the DISCERN Measurement Tool by a faculty member from the Department of Endocrinology and Metabolic Diseases, three faculty members from the Faculty of Nursing, three Diabetes Education Nurses, and a faculty member from the Department of Nutrition and Dietetics. The researcher will introduce the website to adolescents by explaining its name and how to use it. Individuals in the intervention group will also be given usernames and passwords to access the site. New topics, blog posts, and quizzes related to the topic will be added to the site each week, and a reminder message will be sent to individuals in the intervention group when a new topic is added. The website will include an interface where members can log in to their own pages, enter blood glucose measurements, access training modules, exchange messages, and perform administrative tasks (user lists, monitoring all measurements, and tracking training results). The "Contact" page on the website will allow users to send messages to site administrators. Six menus are planned for the website: "Home", "Our Team", "Blog", "Training", "Surveys", and "Contact". Blog Menu: This will be a space where members can chat with each other and share their experiences. The aim is to encourage members to comment on topics determined by the site administrator and share their experiences. After using the website, everyone will be given the opportunity to comment on the materials provided. Educational materials cover topics such as Type 1 diabetes, nutrition for young people with diabetes, carbohydrate counting, acute complications such as hypoglycemia, long-term complications, physical exercise in diabetes, diabetes treatment, insulin, and continuous glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

* T1DM adolescents and their mothers who have internet access at home,
* have a DEPS-R score of 20 or higher,
* are between the ages of 12 and 18,
* have been diagnosed with T1DM at least one year ago,
* have no other chronic illness other than T1DM, and
* agree to participate in the study

Exclusion Criteria:

* Diabetes diagnosis lasted less than one year.
* The adolescent has a chronic condition other than T1DM.
* The adolescent and their mother have cognitive or perceptual disabilities in understanding the website's content.
* Participants who did not complete the training program.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Adolescents with Type 1 DM who participated in the web-based training program experienced a decrease in their disordered eating behavior symptom scores. | AFTER 6 MONTHS
  The Diabetes Eating Disorders Questionnaire and the Dutch Eating Behavior Questionnaire will be used to assess disordered eating behavior. Measurements are planned to be taken at baseline (T0), 1 month (T1), 3 months (T2), and 6 months (T3) time points before the program. A change of at least 20% in the relevant scale scores between T0 and T3, or a statistically significant change with p<0.05, is defined as the success criterion.

SECONDARY OUTCOMES:
Decrease in HbA1c values of adolescents with Type 1 DM who participated in the web-based education program. | AFTER 6 MONTHS
  HbA1c laboratory results will be evaluated at time points T0 (baseline), T2 (3 months), and T3 (6 months). A change of at least 0.5 points in mean HbA1c compared to baseline or a significant change (p<0.05) in the percentage of achieving a clinically significant target (e.g., ≤7.5% as defined by the study) was defined as the success criterion.
Decrease in diabetes self-management skills scores (T1DDYÖS) of adolescents with Type 1 DM who participated in the web-based education program. | AFTER 6 MONTHS
  The T1DDYÖÖ scale will be evaluated at time points T0, T1, and T3 (6 months). A change of at least 15% in scale scores from T0 to T3, or a statistically significant change with p<0.05, is defined as the success criterion.

IPD SHARING:
Plan to Share IPD: Undecided
I don't have detailed information on this subject. Therefore, I'm undecided at the moment.

REFERENCES:
- [Result] Pinsker JE, Nguyen C, Young S, Fredericks GJ, Chan D. A pilot project for improving paediatric diabetes outcomes using a website: the Pediatric Diabetes Education Portal. J Telemed Telecare. 2011;17(5):226-30. doi: 10.1258/jtt.2010.100812. Epub 2011 May 12. PMID 21565846
- [Result] Couch R, Jetha M, Dryden DM, Hooten N, Liang Y, Durec T, Sumamo E, Spooner C, Milne A, O'Gorman K, Klassen TP. Diabetes education for children with type 1 diabetes mellitus and their families. Evid Rep Technol Assess (Full Rep). 2008 Apr;(166):1-144. PMID 18620470
- [Result] Lowes L, Eddy D, Channon S, McNamara R, Robling M, Gregory JW; DEPICTED study team. The experience of living with type 1 diabetes and attending clinic from the perception of children, adolescents and carers: analysis of qualitative data from the DEPICTED study. J Pediatr Nurs. 2015 Jan-Feb;30(1):54-62. doi: 10.1016/j.pedn.2014.09.006. Epub 2014 Sep 28. PMID 25308399
- [Result] Polfuss M, Babler E, Bush LL, Sawin K. Family Perspectives of Components of a Diabetes Transition Program. J Pediatr Nurs. 2015 Sep-Oct;30(5):748-56. doi: 10.1016/j.pedn.2015.05.010. Epub 2015 Jun 15. PMID 26088279
- [Result] Shiel EV, Hemingway S, Burton K, King N. Self-management of type 1 diabetes in young adults: Is it impeded by aspects of everyday life? A scoping review. Diabetes Metab Syndr. 2023 Dec;17(12):102918. doi: 10.1016/j.dsx.2023.102918. Epub 2023 Nov 30. PMID 38064953
- See also: The Diabetes Atlas — https://diabetesatlas.org/
- See also: American Diabetes Association — https://diabetes.org/
- Available data/document: Individual Participant Data Set: The Diabetes Eating Problems — http://jeyned.com — Statistically significant change with p<0.05 was determined as the success criterion.p<0.05 was determined as the success cr